CLINICAL TRIAL: NCT01928615
Title: LISAH: An Open-label, Randomised Phase II Study Assessing Quality of Life Associated With Subcutaneous Trastuzumab Injected Into the Thigh or Upper Arm in Patients With HER2-positive Early Breast Cancer
Brief Title: A Study of Subcutaneously Administered Herceptin (Trastuzumab) in Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Early Breast Cancer
Acronym: LISAH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Problems with drug supply
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML28786; 2013-001023-39 (EudraCT Number)
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Drug Therapy

ARMS (2):
- Trastuzumab - Thigh first, then upper arm (Experimental): In the run-in phase, participants received trastuzumab intravenously every 3 weeks for 18 weeks (Cycles 1-6). They first received trastuzumab 8 mg/kg once (Cycle 1) followed by trastuzumab 6 mg/kg 5 times for 15 weeks (Cycles 2-6). Participants could also receive a maximum of 6 cycles of standard chemotherapy for early breast cancer (neo-adjuvant or adjuvant) in the run-in phase. Following the run-in phase, participants received trastuzumab 600 mg subcutaneously (SC) every 3 weeks into the thigh for 12 weeks (Cycles 7-10) followed by trastuzumab 600 mg SC every 3 weeks into the upper arm for 12 weeks (Cycles 11-14). In Cycles 15-18, participants received trastuzumab 600 mg SC every 3 weeks into either the thigh or the upper arm (participant's choice) for 12 weeks (Cycles 15-18).
  Interventions: Drug: Trastuzumab - intravenous solution; Drug: Trastuzumab - subcutaneous solution; Drug: Chemotherapy
- Trastuzumab - Upper arm first, then thigh (Experimental): In the run-in phase, participants received trastuzumab intravenously every 3 weeks for 18 weeks (Cycles 1-6). They first received trastuzumab 8 mg/kg once (Cycle 1) followed by trastuzumab 6 mg/kg 5 times for 15 weeks (Cycles 2-6). Participants could also receive a maximum of 6 cycles of standard chemotherapy for early breast cancer (neo-adjuvant or adjuvant) in the run-in phase. Following the run-in phase, participants received trastuzumab 600 mg subcutaneously (SC) every 3 weeks into the upper arm for 12 weeks (Cycles 7-10) followed by trastuzumab 600 mg SC every 3 weeks into the thigh for 12 weeks (Cycles 11-14). In Cycles 15-18, participants received trastuzumab 600 mg SC every 3 weeks into either the thigh or the upper arm (participant's choice) for 12 weeks (Cycles 15-18).
  Interventions: Drug: Trastuzumab - intravenous solution; Drug: Trastuzumab - subcutaneous solution; Drug: Chemotherapy

INTERVENTIONS:
Drug: Trastuzumab - intravenous solution — Trastuzumab was supplied as a powder to be reconstituted as a solution for intravenous infusion.
  Other Names: Herceptin; Ro 45-2317
Drug: Trastuzumab - subcutaneous solution — Trastuzumab was supplied as a solution for subcutaneous injection.
  Other Names: Herceptin; Ro 45-2317
Drug: Chemotherapy — Standard chemotherapy for early breast cancer.

SUMMARY:
This open-label, randomized crossover study evaluated the quality of life, efficacy, and safety of subcutaneous Herceptin (trastuzumab) injected either into the thigh or the upper arm of participants with early HER2-positive breast cancer.

DETAILED DESCRIPTION:
In the run-in phase, participants received trastuzumab intravenously every 3 weeks for 18 weeks (Cycles 1-6). They first received trastuzumab 8 mg/kg once (Cycle 1) followed by trastuzumab 6 mg/kg 5 times for 15 weeks (Cycles 2-6). Participants could also receive a maximum of 6 cycles of standard chemotherapy for early breast cancer (neo-adjuvant or adjuvant) in the run-in phase.

Following the run-in phase, participants were randomized to receive trastuzumab 600 mg subcutaneously every 3 weeks in the thigh and upper arm in a cross-over design for a total of 24 weeks (Cycles 7-14). They received trastuzumab either in the thigh first for 4 cycles (Cycles 7-10) followed by trastuzumab in the upper arm for 4 cycles (Cycles 11-14) or the upper arm first (Cycles 7-10) followed by the thigh (Cycles 11-14). For Cycles 15-18, participants could choose the injection site for trastuzumab 600 mg subcutaneously every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ years of age.
* HER2-positive early breast cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Hormonal therapy will be allowed as per institutional guidelines.
* Patients must be Herceptin (trastuzumab) naïve.
* Left ventricular ejection fraction (LVEF) of ≥ 55%.
* Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast.
* No evidence of residual, locally recurrent, or metastatic disease after completion of surgery and chemotherapy, or during concurrent chemotherapy (neo-adjuvant or adjuvant).
* Use of concurrent curative radiotherapy will be permitted.

Exclusion Criteria:

* History of other malignancy which could affect compliance with the protocol or interpretation of results. Patients with curatively treated carcinoma in situ of the cervix or basal cell carcinoma, and patients with other curatively treated malignancies who have been disease-free for at least 5 years, are eligible.
* Patients with severe dyspnea at rest or requiring supplementary oxygen therapy.
* Patients with other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness.
* Serious cardiac illness or medical conditions that would preclude the use of Herceptin, specifically, a history of documented congestive heart failure (CHF), high-risk uncontrolled arrhythmias, angina pectoris requiring medication, clinically significant valvular disease, evidence of transmural infarction on electrocardiogram (ECG), or diagnosed poorly controlled hypertension.
* Pregnant or lactating women.
* Women of childbearing potential and male patients with partners of childbearing potential who are unable or unwilling to use adequate contraceptive measures during study treatment.
* Concurrent enrollment in another clinical trial using an investigational anti-cancer treatment, including hormonal therapy, bisphosphonate therapy, and immunotherapy, within 28 days prior to the first dose of study treatment.
* Known hypersensitivity to trastuzumab, murine proteins, to any of the excipients of Herceptin including hyaluronidase, or a history of severe allergic or immunological reactions, eg, difficult to control asthma.
* Inadequate bone marrow, hepatic, or renal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Austria (2):
  - Innsbruck
  - Salzburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Neither of the 2 enrolled participants were randomized to 1 of the 2 crossover treatment arms. Randomization would not have occurred until after Cycle 6. Both participants only received 1 cycle of treatment.
Groups:
- Trastuzumab: In the run-in phase, participants received trastuzumab intravenously every 3 weeks for 18 weeks (Cycles 1-6). They first received trastuzumab 8 mg/kg once (Cycle 1) followed by trastuzumab 6 mg/kg 5 times for 15 weeks (Cycles 2-6). Following the run-in phase, participants were randomized to receive trastuzumab 600 mg subcutaneously every 3 weeks in the thigh and upper arm in a cross-over design for a total of 24 weeks (Cycles 7-14). They received trastuzumab either in the thigh first for 4 cycles (Cycles 7-10) followed by trastuzumab in the upper arm for 4 cycles (Cycles 11-14) or the upper arm first (Cycles 7-10) followed by the thigh (Cycles 11-14). In Cycles 15-18, participants received trastuzumab 600 mg SC every 3 weeks into either the thigh or the upper arm (participant's choice) for 12 weeks (Cycles 15-18).
Period: Overall Study
Arm/Group | Trastuzumab
Started | 2
Completed | 0
Not Completed | 2
Not completed — Study Terminated by Sponsor | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set: All participants who were enrolled in the study.
Arm/Group | Trastuzumab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Score
Description: Participants rated their quality of life on a visual analog scale (VAS) at the end of each cycle for Cycles 7-14. The left-end of the VAS represented the lowest-rated quality of life and the right-end of the VAS represented the highest-rated quality of life. Both the mean ratings for injections into the thigh and the upper arm and the minimum ratings for during injections into the thigh and the upper arm are reported. Quality of life scores ranged from 1 to 100 with a higher score indicating a better rated quality of life.
Time Frame: Cycles 7-14 (Weeks 19-42, 24 weeks total)
Population: Modified intent-to-treat population: All participants who received at least 1 dose of study medication and who have at least 1 quality of life score in each treatment period (Cycles 7-10 and Cycle 11-14).
  Due to the low enrollment (n = 2) and premature termination of the study, the Outcome Measure was not analyzed.
Groups:
- Trastuzumab - Thigh First, Then Upper Arm: In the run-in phase, participants received trastuzumab intravenously every 3 weeks for 18 weeks (Cycles 1-6). They first received trastuzumab 8 mg/kg once (Cycle 1) followed by trastuzumab 6 mg/kg 5 times for 15 weeks (Cycles 2-6). Following the run-in phase, participants received trastuzumab 600 mg subcutaneously (SC) every 3 weeks into the thigh for 12 weeks (Cycles 7-10) followed by trastuzumab 600 mg SC every 3 weeks into the upper arm for 12 weeks (Cycles 11-14). In Cycles 15-18, participants received trastuzumab 600 mg SC every 3 weeks into either the thigh or the upper arm (participant's choice) for 12 weeks (Cycles 15-18).
- Trastuzumab - Upper Arm First, Then Thigh: In the run-in phase, participants received trastuzumab intravenously every 3 weeks for 18 weeks (Cycles 1-6). They first received trastuzumab 8 mg/kg once (Cycle 1) followed by trastuzumab 6 mg/kg 5 times for 15 weeks (Cycles 2-6). Following the run-in phase, participants received trastuzumab 600 mg subcutaneously (SC) every 3 weeks into the upper arm for 12 weeks (Cycles 7-10) followed by trastuzumab 600 mg SC every 3 weeks into the thigh for 12 weeks (Cycles 11-14). In Cycles 15-18, participants received trastuzumab 600 mg SC every 3 weeks into either the thigh or the upper arm (participant's choice) for 12 weeks (Cycles 15-18).
Arm/Group | Trastuzumab - Thigh First, Then Upper Arm | Trastuzumab - Upper Arm First, Then Thigh
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from Baseline to death from any cause.
Time Frame: Baseline to the end of the study (up to 54 weeks)
Population: Intent-to-treat population: All participants who received at least 1 dose of study medication.
  Due to the low enrollment (n = 2) and premature termination of the study, the Outcome Measure was not analyzed.
Arm/Group | Trastuzumab - Thigh First, Then Upper Arm | Trastuzumab - Upper Arm First, Then Thigh
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Disease-free Survival
Description: Disease-free survival was defined as the time in months from Baseline to disease recurrence or death, whichever occurred first.
Time Frame: Baseline to the end of the study (up to 54 weeks)
Population: as for outcome 2
Arm/Group | Trastuzumab - Thigh First, Then Upper Arm | Trastuzumab - Upper Arm First, Then Thigh
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Health Care Provider's Satisfaction With the Injection Site
Description: The health care provider for each participant was asked to rate their satisfaction with the 2 injection sites, thigh and upper arm, on a scale of 1 to 10, where 10 represents greater satisfaction. Ratings were made at the end of Cycles 10 and 14.
Time Frame: End of Cycles 10 and 14 (Weeks 30 and 42)
Population: as for outcome 2
Arm/Group | Trastuzumab - Thigh First, Then Upper Arm | Trastuzumab - Upper Arm First, Then Thigh
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Participant's Satisfaction With the Injection Site
Description: Each participant was asked to rate their satisfaction with the 2 injection sites, thigh and upper arm, on a scale of 1 to 10, where 10 represents greater satisfaction. Ratings were made at the end of Cycles 10 and 14.
Time Frame: End of Cycles 10 and 14 (Weeks 30 and 42)
Population: as for outcome 2
Arm/Group | Trastuzumab - Thigh First, Then Upper Arm | Trastuzumab - Upper Arm First, Then Thigh
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Preferring Each Injection Site
Description: Participants were asked which of the 2 injection sites was their preferred site at the end of Cycle 14.
Time Frame: End of Cycle 14 (Week 42)
Population: as for outcome 2
Arm/Group | Trastuzumab - Thigh First, Then Upper Arm | Trastuzumab - Upper Arm First, Then Thigh
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Intent-to-treat population: All participants who received at least 1 dose of study medication.
Arm/Group | Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=2)
Common cold (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.